CLINICAL TRIAL: NCT01320579
Title: Phase II Study to Investigate the Properties of Topical Twice Daily Doses of 2.5% and 5% Cis-urocanic Acid in Comparison to Active Comparator 0.1% Protopic® for up to 28 Days in Patients With Moderate or Severe Atopic Dermatitis
Brief Title: Investigation of the Efficacy of 2.5% and 5% Cis-urocanic Acid in Patients With Moderate or Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioCis Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL09002; 2010-023543-15 (EudraCT Number)
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; cis-urocanic acid
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Tacrolimus; Ointments

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 2 Cis-UCA 5% emulsion cream (Experimental)
  Interventions: Drug: Cis-UCA 5% emulsion cream
- Group 3 Placebo cis-UCA emulsion cream (Placebo Comparator)
  Interventions: Drug: Placebo for cis-UCA emulsion cream
- Group 4 Protopic® 0.1% ointment (Active Comparator)
  Interventions: Drug: Protopic® 0.1% ointment
- Group 1 Cis-UCA 2.5% emulsion cream (Experimental)
  Interventions: Drug: Cis-UCA 2.5% emulsion cream

INTERVENTIONS:
Drug: Cis-UCA 2.5% emulsion cream — 2.5% cis-UCA in emulsion cream base twice daily, amount of a fingertip per one hand (i.e. palm + thumb + fingers) area, applied topically as a thin layer on the affected skin area of approximate size of maximally three hand areas for up to 28 days (one fingertip per one hand area)
  Other Names: Cis-UCA 2.5%
  Arms: Group 1 Cis-UCA 2.5% emulsion cream
Drug: Cis-UCA 5% emulsion cream — 5% cis-UCA in emulsion cream base twice daily, amount of a fingertip per one hand (i.e. palm + thumb + fingers) area, applied topically as a thin layer on the affected skin area of approximate size of maximally three hand areas for up to 28 days (one fingertip per one hand area)
  Other Names: Cis-UCA 5%
  Arms: Group 2 Cis-UCA 5% emulsion cream
Drug: Placebo for cis-UCA emulsion cream — The placebo for cis-UCA product (emulsion cream base) twice daily, amount of a fingertip per one hand area applied topically as a thin layer on the affected skin area on of approximate size of maximally three hand areas for up to 28 days (one fingertip per one hand area).
  Other Names: Placebo
  Arms: Group 3 Placebo cis-UCA emulsion cream
Drug: Protopic® 0.1% ointment — 0.1% Protopic® twice daily, amount of a fingertip per one hand area applied topically as a thin layer on the affected skin area of approximate size of maximally three hand areas for up to 28 days (one fingertip per one hand area).
  Other Names: Protopic®
  Arms: Group 4 Protopic® 0.1% ointment

SUMMARY:
The purpose of this study is to evaluate dose response, safety, tolerability and efficacy of 2.5% and 5% cis-UCA in comparison to placebo and active comparator in the treatment of adult patients with moderate or severe chronic atopic dermatitis.

DETAILED DESCRIPTION:
This is a Phase II multi-centre, double-blinded, vehicle-controlled, repeated and multiple dose, study to evaluate dose response, safety, tolerability and efficacy of 2.5% and 5% cis-UCA compared to placebo, and investigator-blinded to compare the safety, tolerability and efficacy of cis-UCA to the active comparator Protopic® 0.1% in patients with moderate or severe chronic atopic dermatitis treated for up to 28 days.

The primary objective is to compare the efficacy of two different doses of cis-UCA (2.5% and 5%) with placebo for up to 28 days in adult patients with moderate or severe chronic atopic dermatitis to determine the dose of cis-UCA for further clinical development.

Secondary objectives are as follows:

* To evaluate safety and tolerability of cis-UCA after topical twice daily doses of 2.5% and 5% for up to 28 days in adult patients with moderate or severe chronic atopic dermatitis.
* To evaluate dose response after topical twice daily doses of 2.5% and 5% for up to 28 days in adult subjects with moderate or severe chronic atopic dermatitis.
* To compare the efficacy and safety of 2.5% and 5% of cis-UCA to the efficacy and safety of 0.1% Protopic® after topical twice daily doses for up to 28 days in adult patients with moderate or severe chronic atopic dermatitis

The key eligibility criteria are the following: patients with moderate or severe chronic atopic dermatitis, at least 18 years of age, with no current treatment for atopic dermatitis with active systemic medication or active topical treatment in the planned investigational area, and with no history of any significant disease that would affect the use of cis-UCA or comparator.

In total, up to 150 adult patients (both males and females; at least 20% of each gender) with moderate or severe chronic atopic dermatitis will be included in the study. Up to 36 adult patients (both males and females) will be included in each treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained prior to any screening procedure
* Caucasian male or female patient
* At least 18 years of age
* Weight at least 45 kg
* Patient with moderate or severe chronic atopic dermatitis
* Good general health ascertained by medical history, physical examination and laboratory determinations, showing no signs of clinically significant findings, except chronic atopic dermatitis
* Negative pregnancy test (premenopausal female patient) at screening and use of adequate contraceptive measures (both male and female patients) throughout the study and 30 days after the last cis-UCA dose

Exclusion Criteria:

* History of other significant skin disease, or skin manifestations of allergic illness or other dermatologic condition, except chronic moderate or severe atopic dermatitis, that would interfere with the trial assessments or compromise the patient's safety according to the opinion of the Investigator
* Present symptoms of other skin diseases, except chronic atopic dermatitis, that could disturb the study assessment and evaluation of the skin
* Current use of any active systemic medication for chronic atopic dermatitis within one month
* Current use of active topical medication in the planned investigational area for chronic atopic dermatitis within two weeks
* History of a sunny holiday, UV-light therapy or solarium use within one month before beginning of study treatments, or planning such during the study or within 7 days after the study
* Allergy to cis-UCA, or any constituents of the placebo emulsion cream or any constituents of Protopic® ointment
* History of any skin-related cancer
* Congenital or acquired immunodeficiency or ongoing therapy that cause immunosuppression
* Earlier participation in a clinical study performed with cis-UCA
* Any clinically significant laboratory test result
* Suspected current drug or alcohol abuse
* Clinically significant illness during the 4 weeks prior to the first dose administration
* Any other condition that in the opinion of the Investigator would interfere with the evaluation of the study results or constitute a health hazard for the patient
* Unwillingness or doubtful capacity to comply with the protocol
* Doubtful availability to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Clinical Skin Assessment of erythema, oedema/papulation, oozing/crusts, excoriations, and lichenification | 37 days

SECONDARY OUTCOMES:
Skin Erythema measurement | 37 days
Transepidermal Water Loss (TEWL) measurement | 37 days
Visual Analogue Scale (VAS) assessment for itching (pruritus) of the treatment area | 37 days
Physician Global Assessment (PGA) | 37 days

CONTACTS AND LOCATIONS:
Overall Officials: Sakari Reitamo, Professor, Principal Investigator — Helsinki University Central Hospital, Skin and Allergy Hospital
Locations (7):
- Finland (7):
  - Helsinki University Central Hospital, Skin and Allergy Hospital, Helsinki
  - Mehiläinen Medical Center Kuopio, Kuopio
  - Lohja Hospital, Clinic of Dermatology and Allergology, Lohja
  - FinnMedi Oy, Tampere
  - Mehiläinen Medical Center Turku, Turku
  - Pulssi Medical Center, Turku
  - Turku University Hospital, Department of Dermatology and Venereal Diseases, Turku

REFERENCES:
- [Background] Bieber T. Atopic dermatitis. N Engl J Med. 2008 Apr 3;358(14):1483-94. doi: 10.1056/NEJMra074081. No abstract available. PMID 18385500
- [Background] Cork MJ, Danby SG, Vasilopoulos Y, Hadgraft J, Lane ME, Moustafa M, Guy RH, Macgowan AL, Tazi-Ahnini R, Ward SJ. Epidermal barrier dysfunction in atopic dermatitis. J Invest Dermatol. 2009 Aug;129(8):1892-908. doi: 10.1038/jid.2009.133. Epub 2009 Jun 4. PMID 19494826
- [Background] De Fabo EC, Noonan FP. Mechanism of immune suppression by ultraviolet irradiation in vivo. I. Evidence for the existence of a unique photoreceptor in skin and its role in photoimmunology. J Exp Med. 1983 Jul 1;158(1):84-98. doi: 10.1084/jem.158.1.84. PMID 6223114
- [Background] Severity scoring of atopic dermatitis: the SCORAD index. Consensus Report of the European Task Force on Atopic Dermatitis. Dermatology. 1993;186(1):23-31. doi: 10.1159/000247298. PMID 8435513
- [Background] Hanifin JM, Reed ML; Eczema Prevalence and Impact Working Group. A population-based survey of eczema prevalence in the United States. Dermatitis. 2007 Jun;18(2):82-91. doi: 10.2310/6620.2007.06034. PMID 17498413
- [Background] Rajka G, Langeland T. Grading of the severity of atopic dermatitis. Acta Derm Venereol Suppl (Stockh). 1989;144:13-4. doi: 10.2340/000155551441314. PMID 2800895
- [Background] Wolkerstorfer A, de Waard van der Spek FB, Glazenburg EJ, Mulder PG, Oranje AP. Scoring the severity of atopic dermatitis: three item severity score as a rough system for daily practice and as a pre-screening tool for studies. Acta Derm Venereol. 1999 Sep;79(5):356-9. doi: 10.1080/000155599750010256. PMID 10494710
- [Derived] Peltonen JM, Pylkkanen L, Jansen CT, Volanen I, Lehtinen T, Laihia JK, Leino L. Three randomised phase I/IIa trials of 5% cis-urocanic acid emulsion cream in healthy adult subjects and in patients with atopic dermatitis. Acta Derm Venereol. 2014 Jul;94(4):415-20. doi: 10.2340/00015555-1735. PMID 24284985